CLINICAL TRIAL: NCT04654416
Title: Clinical Outcome of Patients With COVID-19 Pneumonia Treated With Corticosteroids and Colchicine in Colombia
Brief Title: Clinical Outcome of Patients With COVID-19 Pneumonia Treated With Corticosteroids and Colchicine
Status: Completed | Type: Observational
Sponsor: Clínica Medellín - Grupo Quirónsalud (Other)
Responsible Party: Principal Investigator, Miguel Alejandro Pinzón, Internal Medicine - Infectious Diseases Specialist, Clínica Medellín - Grupo Quirónsalud
Other Study IDs: 04-2020
Record Dates: First submitted 2020-12-02; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Covid-19
Keywords: Dexamethasone; Corticosteroid; Covid-19; Pneumonia; Colchicine; Clinical outcome
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — Adrenal Cortex Hormones; Colchicine

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Steroids: Dexamethasone 6mg intravenous OD for seven to ten days
  Interventions: Drug: Corticosteroid with or without colchicine
- Colchicine: Patients treated with colchicine at a dose of 0.5 mg every 12 hours for 7 to 14 days.
  Interventions: Drug: Corticosteroid with or without colchicine

INTERVENTIONS:
Drug: Corticosteroid with or without colchicine — We describe the clinical outcome of patients treated with corticosteroid and colchicine

SUMMARY:
Cross sectional study of 301 adult patients with Covid-19 Pneumonia treated with corticosteroid and/or colchicine

DETAILED DESCRIPTION:
A cross sectional study of 301 adult patients with Covid-19 Pneumonia confirmed by Real-Time Polymerase Chain Reaction for SARS-CoV2 (RT-PCR SARS-CoV2), Berlin protocol, who required hospitalization in three hospitals in Antioquia, Colombia. Patients were treated according to the institutional protocol (from March 20, 2020 to June 30, 2020) with corticosteroid if the patient required supplemental oxygen. From July 1, 2020, the management protocol changed with the addition of colchicine to all patients admitted to the institutions. The treatment was supervised and monitored by the same specialist in infectology of the institutions.

We describe the clinical manifestations and outcomes of the patients who received these treatments. The patient's information was analyzed according to the outcome of interest (alive/dead) with univariate, bivariate, and multivariate measures to adjust the variables that presented statistical association.

ELIGIBILITY:
Inclusion Criteria:

* The included patients were older than 18 years hospitalized for Covid-19 Pneumonia, confirmed positive by Real-Time Reverse Transcription Polymerase Chain Reaction for SARS-CoV2 (RT-PCR SARS-Cov2) by Berlin protocol. The samples were taken from a nasopharyngeal swab.
* The patients should also have radiological confirmation of Pneumonia, mostly chest tomography or chest X-rays, to support the diagnosis of Covid-19 Pneumonia.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Covid-19 pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
Outcome | March 20 to August 07, 2020
  Dead or alive

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Medellín - Grupo Quirónsalud, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Mahase E. Coronavirus covid-19 has killed more people than SARS and MERS combined, despite lower case fatality rate. BMJ. 2020 Feb 18;368:m641. doi: 10.1136/bmj.m641. No abstract available. PMID 32071063
- [Background] Yao X, Ye F, Zhang M, Cui C, Huang B, Niu P, Liu X, Zhao L, Dong E, Song C, Zhan S, Lu R, Li H, Tan W, Liu D. In Vitro Antiviral Activity and Projection of Optimized Dosing Design of Hydroxychloroquine for the Treatment of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Clin Infect Dis. 2020 Jul 28;71(15):732-739. doi: 10.1093/cid/ciaa237. PMID 32150618
- [Background] de Wit E, Feldmann F, Cronin J, Jordan R, Okumura A, Thomas T, Scott D, Cihlar T, Feldmann H. Prophylactic and therapeutic remdesivir (GS-5734) treatment in the rhesus macaque model of MERS-CoV infection. Proc Natl Acad Sci U S A. 2020 Mar 24;117(12):6771-6776. doi: 10.1073/pnas.1922083117. Epub 2020 Feb 13. PMID 32054787
- [Background] RECOVERY Collaborative Group; Horby P, Lim WS, Emberson JR, Mafham M, Bell JL, Linsell L, Staplin N, Brightling C, Ustianowski A, Elmahi E, Prudon B, Green C, Felton T, Chadwick D, Rege K, Fegan C, Chappell LC, Faust SN, Jaki T, Jeffery K, Montgomery A, Rowan K, Juszczak E, Baillie JK, Haynes R, Landray MJ. Dexamethasone in Hospitalized Patients with Covid-19. N Engl J Med. 2021 Feb 25;384(8):693-704. doi: 10.1056/NEJMoa2021436. Epub 2020 Jul 17. PMID 32678530
- [Background] Deftereos SG, Giannopoulos G, Vrachatis DA, Siasos GD, Giotaki SG, Gargalianos P, Metallidis S, Sianos G, Baltagiannis S, Panagopoulos P, Dolianitis K, Randou E, Syrigos K, Kotanidou A, Koulouris NG, Milionis H, Sipsas N, Gogos C, Tsoukalas G, Olympios CD, Tsagalou E, Migdalis I, Gerakari S, Angelidis C, Alexopoulos D, Davlouros P, Hahalis G, Kanonidis I, Katritsis D, Kolettis T, Manolis AS, Michalis L, Naka KK, Pyrgakis VN, Toutouzas KP, Triposkiadis F, Tsioufis K, Vavouranakis E, Martinez-Dolz L, Reimers B, Stefanini GG, Cleman M, Goudevenos J, Tsiodras S, Tousoulis D, Iliodromitis E, Mehran R, Dangas G, Stefanadis C; GRECCO-19 investigators. Effect of Colchicine vs Standard Care on Cardiac and Inflammatory Biomarkers and Clinical Outcomes in Patients Hospitalized With Coronavirus Disease 2019: The GRECCO-19 Randomized Clinical Trial. JAMA Netw Open. 2020 Jun 1;3(6):e2013136. doi: 10.1001/jamanetworkopen.2020.13136. PMID 32579195
- [Background] Dong L, Hu S, Gao J. Discovering drugs to treat coronavirus disease 2019 (COVID-19). Drug Discov Ther. 2020;14(1):58-60. doi: 10.5582/ddt.2020.01012. PMID 32147628
- [Background] Russell CD, Millar JE, Baillie JK. Clinical evidence does not support corticosteroid treatment for 2019-nCoV lung injury. Lancet. 2020 Feb 15;395(10223):473-475. doi: 10.1016/S0140-6736(20)30317-2. Epub 2020 Feb 7. No abstract available. PMID 32043983
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578